CLINICAL TRIAL: NCT07020117
Title: NECTINIUM-2: A Phase 1b, 2 Part, Multicenter, Single Arm, Open Label Study to Evaluate the Safety and Efficacy of a Nectin-4 Radiopharmaceutical ([225Ac]Ac-AKY-1189) in Patients With Previously Treated Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study of [225Ac]Ac-AKY-1189 in Patients With Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Aktis Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AKY-1189-01
Record Dates: First submitted 2025-05-28; First posted 2025-06-13 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Urothelial Carcinoma Bladder; Triple Negative Breast Cancer (TNBC); Hormone Receptor Positive Breast Adenocarcinoma; Non Small Cell Lung Cancer; Cervical Adenocarcinoma; Colorectal Adenocarcinoma; Head and Neck Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Head and Neck Neoplasms | interventions — Therapeutics; X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [225Ac]Ac-AKY-1189 (Experimental)
  Interventions: Drug: [225Ac]Ac-AKY-1189 (therapeutic); Drug: [64Cu]Cu-AKY-1189 (imaging)

INTERVENTIONS:
Drug: [225Ac]Ac-AKY-1189 (therapeutic) — [225Ac]Ac-AKY-1189 Injection
Drug: [64Cu]Cu-AKY-1189 (imaging) — [64Cu]Cu-AKY-1189 Injection

SUMMARY:
This is a first-in-human Phase 1b, 2-part, multicenter open-label clinical study to evaluate safety and efficacy of a Nectin-4 radiopharmaceutical ([225Ac]Ac-AKY-1189) in patients with locally advanced or metastatic solid tumors and to establish the maximum tolerated dose (MTD) or maximum administered dose (MAD) and the recommended Phase 2 dose.

DETAILED DESCRIPTION:
This study consists of two parts (Part 1 and 2).

Part 1 is the dose escalation portion of the study, which will investigate ascending doses of [225Ac]Ac-AKY-1189 (up to 6 cycles) in patients with locally advanced or metastatic solid tumors. The aim of Part 1 is to determine the maximum tolerated dose (MTD) or maximum administered dose (MAD) and the recommended Phase 2 dose.

Part 2 will be the dose expansion portion of the study and will enroll locally advanced or metastatic solid tumor patients who are identified as Nectin-4 positive by [64Cu] Cu-AKY-1189. Part 2 aims to further assess the efficacy of [225Ac]Ac-AKY-1189 at the RP2D in 3 different cohorts of patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic confirmation of locally advance or metastatic disease
* Radiologic confirmation on CT of at least one measurable tumor lesion per RECIST v1.1
* ECOG Performance Status of 0 or 1
* Adequate end-organ function
* Ability to give informed consent and comply with study requirements
* Patients with CNS metastases are eligible if they have received therapy and are neurologically stable, asymptomatic and not receiving corticosteroids
* Documented disease progression on prior line of therapy for metastatic disease

Exclusion Criteria:

* Prior treatment with a therapeutic radiopharmaceutical
* Prior treatment with a Nectin-4 targeted therapy, except enfortumab vedotin
* Received an investigational agent within the previous 28days
* Prior treatment with a cytotoxic chemotherapy, targeted therapy, biologic agent, immunotherapy or external-beam radiotherapy in the 3 weeks prior to study treatment
* Concurrent serious medical condition that would impair study participation or impact the assessment of treatment related toxicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-08-22 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2032-06 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Patients with Dose-Limiting Toxicities | From enrollment to the end of Cycle 1 (each cycle is 28 days)
  • Dose-limiting toxicities (DLTs) is defined as any predefined AE occurring during the DLT observation period, except those that are clearly and incontrovertibly due to extraneous circumstances. The number of patients who experience a DLT in Part 1, will be reported by dose level.
Part 1: Occurence of Adverse Events by Severity | Up to the End of Treatment (30 days after the last dose)
  • An AE is defined as any untoward medical occurrence in a participant administered study drug, which does not necessarily have to have a causal relationship with the study drug. The number of patients experiencing an AE in Part 1 will be reported.
Part 2: Objective Response Rate (ORR) | Up to 30 days following last administration
  • Objective response rate is defined as the percentage of patients who achieved a best overall response of confirmed Complete Response (CR) or Partial Response (PR), as determined by the investigator based on RECIST 1.1, by tumor types.

SECONDARY OUTCOMES:
Part 1: Objective Response Rate (ORR) | Up to 30 days following last adminstration
  • Objective response rate is defined as the percentage of patients who achieved a best overall response of confirmed Complete Response (CR) or Partial Response (PR), as determined by the investigator based on RECIST 1.1, by dose level.
Part 2: Occurence of Adverse Events by Severity | Up to End of Treatment (30 days after the last dose)
  • An AE is defined as any untoward medical occurrence in a participant administered study drug, which does not necessarily have to have a causal relationship with the study drug. The number of patients experiencing an AE in Part 2 will be reported.
Part 1 and 2: Duration of Response (DOR) | Up to 5 years after first administration
  • Duration of Response (DoR) was defined as the time from the date of the first documentation of objective response (complete response [CR] or partial response [PR]) to the date of the first objective documentation of progressive disease (PD) or death due to any cause.
Part 1 and 2: Progression-Free Survival (PFS) | Up to 5 years after first administration
  • PFS is defined as the time from treatment initiation to the first documented disease progression per RECIST 1.1 or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - City of Hope, Duarte, California
  - Hoag Memorial Hospital Presbyterian, Irvine, California
  - Biogenix Molecular, LLC, Miami, Florida
  - University of Iowa, Iowa City, Iowa
  - BAMF Health, Grand Rapids, Michigan
  - Icahn School of Medicine at Mt. Sinai, New York, New York
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided